CLINICAL TRIAL: NCT00001154
Title: Lipoprotein Metabolism in Normal Volunteers and Hyperlipoproteinemic Patients
Brief Title: Lipoprotein Metabolism in Normal Volunteers and Patients With High Levels of Lipoproteins
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 760051; 76-H-0051
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-06-23

CONDITIONS: Hypolipoproteinemia; Hypercholesterolemia; Dyslipidemia; Hyperlipidemia
Keywords: Metabolism; HDL; Cholesterol; LDL; Hypoalphalipoproteinemia; Natural History
MeSH Terms: conditions — Hypolipoproteinemias; Hypercholesterolemia; Dyslipidemias; Hyperlipidemias; Hypoalphalipoproteinemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Subjects with new and undefined dyslipidemia

SUMMARY:
Researchers plan to study the fat-rich particles, called lipoproteins, which circulate in the blood. This study is designed to improve understanding of normal, as well as abnormal, lipoprotein metabolism and the role it plays in the development of hardening of the arteries (atherosclerosis).

Patients participating in this study will receive injections of lipoproteins or apolipoproteins (the protein component of lipoproteins) that have been isolated and purified. These lipoproteins will be labeled with small amounts of radioactive material and sterilized before they are injected into the patient.

Patients participating in the study will be required to have blood samples taken, and provide urine samples throughout the course of the study. In addition, patient will be required to follow a specially formulated diet. Patients will be weighed throughout the course of the study.

DETAILED DESCRIPTION:
We propose to investigate human in vivo lipoprotein metabolism using radiolabeled apolipoproteins on plasma lipoproteins. Paired kinetic studies using dual-labeled iodinated lipoproteins and apolipoproteins are performed in healthy volunteer controls with normal lipids and subjects with dyslipidemia under controlled metabolic conditions. Studies are designed to formulate metabolic pathways in patients with undefined genetic disorders of lipid metabolism as well as in healthy volunteers to provide original insights into normal and pathologic metabolic pathways. All kinetic data is computer analyzed to provide quantitative data and facilitate direct comparison of multiple studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects with new and undefined dyslipidemia-particularly familial disorders with extreme phenotypes.

Healthy normal volunteers - (18 years old or older) controls to investigate the formation of HDL for prebeta HDL.

Euthyroid.

EXCLUSION CRITERIA:

Healthy control volunteers are initially screened for secondary causes of hyperlipidemia and are excluded if they have any clinically significant laboratory abnormality (i.e., liver disease, disease, kidney disease, endocrine disease,), chronic medical problems (i.e., hypertension, migraines, inflammatory bowel, hepatitis, HIV) or require any chronic medications (i.e., acne, asthma).

The healthy control volunteers weight must fall within the current guidelines for ideal body weight.

Pregnant women.

Unwilling to follow metabolic diet.

Allergic to iodine.

Unable to sign consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dsylipidemia
Sampling Method: Non-Probability Sample
Enrollment: 759 (Actual)
Dates: Start 1976-09-03 (Actual)

PRIMARY OUTCOMES:
No outcome. This is a disease discover protocol. | 5 years
  Dyslipidemia

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Shamburek, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1976-H-0051.html